CLINICAL TRIAL: NCT02131337
Title: Efficacy Study on Atrial Fibrillation Percutaneous Catheter Ablation With Contact Force Support 2
Brief Title: TactiCath® Prospective Effectiveness Pilot Study
Acronym: EFFICAS II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Collaborators: Endosense (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EFFICAS II Version B
Record Dates: First submitted 2014-04-28; First posted 2014-05-06 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Contact force lesions (Other)
  Interventions: Other: Electrophysiology study

INTERVENTIONS:
Other: Electrophysiology study — after 3 months to check for pulmonary vein isolation (PVI) status

SUMMARY:
EFFICAS II proposes to test the hypothesis that treatment efficacy correlates to contact force parameters applied for pulmonary vein isolation (PVI) during AF ablation.

DETAILED DESCRIPTION:
EFFICAS II is a single-arm, prospective study, where the operator will have access to contact force information and use it actively to optimize the ablation result and adapting power if necessary. The endpoint will correlate contact force parameters initially applied in PV and 3 months PV isolation status, and compare results to those of EFFICAS I.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age but not over 75 years of age
* Patient has at least one episode of sustained (>30s) paroxysmal atrial fibrillation documented by 12-lead ECG, holter monitor, transtelephonic event monitor, telemetry strip, or Pacemaker respectively implantable cardioverter defibrillator (ICD) within 12 months prior to enrolment
* Patient has symptomatic paroxysmal atrial fibrillation (PAF) refractory or intolerant to at least one Class I-IV anti-arrhythmic drug
* Patient is willing and capable of complying with the study protocol requirements, including the specified follow-up scheme
* Patient provides written informed consent prior to enrolment in the study

Exclusion Criteria:

* Not adhering to inclusion criteria
* Active systemic infection
* Recent (within 3 months) cardiac events including myocardial infarction, acute coronary syndrome, percutaneous coronary intervention (PCI), or valve or coronary bypass grafting surgery
* Reversible causes of Arrhythmia including thyroid disorders, acute alcohol intoxication, recent (less than 3 months) major surgical procedures
* Patient has a left atrial diameter > 5.0 cm
* Patient has persistent or long-standing persistent atrial fibrillation (AF)
* Left ventricular ejection fraction < 35%
* New York Heart Association (NYHA) class III or IV
* Previous left atrial heart ablation procedure, either surgical or catheter ablation
* Patient has an intracardiac mural thrombus or has had a ventriculotomy or atriotomy
* Patient has moderate or severe structural heart disease as demonstrated by transthoracic or trans-esophageal echocardiogram of all four chambers of the heart (ventricular dysfunction or valve disease)
* Tricuspid or mitral valve replacement or repair
* If female of childbearing potential - pregnant or breastfeeding
* Patient has a bleeding diathesis or suspected pro-coagulant state
* Patient has contraindication to long-term antithromboembolic therapy (e. g. acetylsalicylic acid, heparin, warfarin)
* Presence of condition that precludes appropriate vascular access
* Heart disease in which corrective surgery is anticipated within 6 months
* Renal failure requiring dialysis
* Patient has a known sensitivity to contrast media (if needed during the procedure) that cannot adequately be controlled with pre-medication (or totally excluded)
* Patient has other anatomic or co-morbid conditions that, in the Investigator's opinion, could limit the patient's ability to participate in the study or to comply with follow-up requirements, or impact the scientific soundness of the study results
* Patient is currently participating in another clinical trial
* Patient is unlikely to survive over one year

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-12; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Number of pulmonary vein isolation (PVI) gaps per vein | 3 months
  Number of gaps in EFFICAS 2 is lower than in EFFICAS 1 and Contact force in EFFICAS 2 has reduced variability than in EFFICAS 1. Confounding parameters such as lesion continuity will be determined for the remaining gaps in EFFICAS 2.

CONTACTS AND LOCATIONS:
Locations (3):
- Czechia (2):
  - IKEM, Prague
  - Na Homolce, Prague
- Asklepios St Georg, Hamburg, Germany